CLINICAL TRIAL: NCT00497731
Title: A Phase I, Open-Label, Multi-Centre Study to Assess the Safety, Tolerability and Pharmacokinetics of AZD1152 Given as a 2 Hour Intravenous Infusion on Two Dose Schedules in Patients With Advanced Solid Malignancies
Brief Title: AZD1152 in Patients With Advanced Solid Malignancies-Study 1
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Efficacy seen in the solid tumour patient population was not sufficient to continue research with AZD1152 monotherapy in solid tumors at that time.
Sponsor: AstraZeneca (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1531C00001
Record Dates: First submitted 2007-07-05; First posted 2007-07-09 (Estimated); Last update posted 2009-06-22 (Estimated); Status verified 2009-06

CONDITIONS: Solid Tumors
Keywords: Advanced solid tumors
MeSH Terms: interventions — 2-((3-((4-((5-(2-((3-fluorophenyl)amino)-2-oxoethyl)-1H-pyrazol-3-yl)amino)quinazolin-7-yl)oxy)propyl)(ethyl)amino)ethyl dihydrogen phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: AZD1152 — 2-hour continuous intravenous infusion

SUMMARY:
The primary purpose of this protocol is to investigate the safety and tolerability of AZD1152 when given as a continuous 2-hour infusion every week and every 2 weeks in patients with advanced solid malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological confirmation of a solid, malignant tumour
* At least measurable or non measurable site of disease as defined by modified RECIST criteria.

Exclusion Criteria:

* Participation in an investigational drug study within 30 days prior to entry or who have not recovered from the effects of an investigational study drug
* Treatment with radiotherapy/chemotherapy with 4 weeks of first dose
* Recent major surgery within 4 weeks prior to entry to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2005-05; Primary Completion 2008-06 (Actual); Study Completion 2009-04 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | Assessed at each visit

SECONDARY OUTCOMES:
Pharmacokinetics | Assessed at predetermined timepoints after dose administration
Effect on biomarkers | Assessed after treatment
Anti-tumor activity | Assessed after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jan Schellens, MD, Principal Investigator — NKI
Locations (2):
- Netherlands (2):
  - Research Site, Amsterdam
  - Research Site, Utrecht